CLINICAL TRIAL: NCT00585299
Title: Effects of Weight Loss on Hepatic and Muscle Lipid Content and on Insulin Sensitivity on Obese Adolescents With NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0212023115; R01HD040787-01 (NIH)
Record Dates: First submitted 2007-12-22; First posted 2008-01-03 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Fatty Liver; Insulin Resistance
Keywords: steatosis; fatty liver; insulin sensitivity; fatty liver (steatosis)
MeSH Terms: conditions — Fatty Liver; Insulin Resistance | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-fat diet (Experimental): 20% kcals from fat diet followed for 8 weeks then 8 weeks of maintenance diet with visits to dietitian every other week
  Interventions: Other: Low-fat diet; Other: Traditional diet
- Traditional (Active Comparator): Traditional low-fat diet given and dietitian follows up in 16 weeks
  Interventions: Other: Traditional diet

INTERVENTIONS:
Other: Low-fat diet — 20% calorie from fat diet followed for 8 weeks then maintenance diet for additional 8 weeks
  Arms: Low-fat diet
Other: Traditional diet — Traditional low-fat diet with dietitian follow-up in 16 weeks

SUMMARY:
To assess whether reversal of fatty liver by moderate weight loss (8% of body weight) will lead to improvements in insulin sensitivity, which will be associated with changes in both glucose status and lipid profiles, in obese children and adolescents with fatty liver who have normal glucose or pre-diabetes.

DETAILED DESCRIPTION:
This study will have two groups: one group that eats a moderate calorie, low-fat diet and is weighed regularly (every other week for 16 weeks) and the other who receives traditional diet therapy and returns in 16 weeks. Both groups will undergo procedures that test glucose tolerance and measure liver and muscle fat content before and after study period.

ELIGIBILITY:
Inclusion Criteria:

* 10 to 21 yrs of age
* Non-smoking
* BMI >95th percentile for age and gender, but BMI <40
* Suspicion of fatty liver, with a high ALT (>35)
* Normal glucose tolerance or prediabetes (impaired glucose tolerance or impaired fasting glucose)

Exclusion Criteria:

* Females of child-bearing potential who are not using birth control
* Pregnant or lactating females
* Current medications except oral anti-diabetic medications and hormonal birth control
* Lipid-lowering medication that increases liver enzymes
* Significant kidney dysfunction (creatinine >1.5 mg/dL)
* Current heavy ethanol use or recent history of binge drinking
* History or evidence of hepatitis A, B, or C, Wilson's Disease, or alpha-1-antitrypsin deficiency
* Known to be HIV positive
* Symptomatic angina pectoris or cardiac insufficiency as defined by the NYHA classification as Functional Class III or IV
* Major vascular event within 6 months of screening (e.g. MI, stroke)
* Active cancer within 5 years prior to screening
* Current systemic disease, including type 1 or 2 diabetes
* Enrolled in another research study within 1 month prior to screening
* Implanted paramagnetic material (all subjects will need to fill out the Yale Magnetic Resonance Center safety checklist)
* Anemia (HCT <35%)

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Liver Enzyme, liver and muscle fat content, glucose tolerance status | 16-18 weeks

SECONDARY OUTCOMES:
plasma lipid levels | 16-18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States